CLINICAL TRIAL: NCT03661736
Title: Growth of Infants With Cow's Milk Allergy Fed an Amino Acid-based Formula Containing Two Human Milk Oligosaccharides: Comparison With World Health Organization (WHO) Growth Standards in an Observational, Single-arm Study
Brief Title: Growth of Infants With Cow's Milk Allergy Fed an Amino Acid-based Formula Containing Two Human Milk Oligosaccharides
Acronym: PLATYPUS
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 17.09.CLI
Record Dates: First submitted 2018-08-22; First posted 2018-09-07 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-08

CONDITIONS: Cow Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Food

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Food for Specific Medical Purpose — Infants aged 1 to 8 months with moderate-to-severe cow's milk allergy fed an amino acid-based formula with two added human milk oligosaccharides

SUMMARY:
The main aim of this study is to provide longitudinal growth data in infants with moderate-to-severe cow's milk allergy fed an amino acid-based formula with two added human milk oligosaccharides.

ELIGIBILITY:
Inclusion Criteria:

1. Full term infant (37 weeks ≤ gestation ≤ 42 weeks)
2. 2500g ≤ birth weight ≤ 4500g
3. Having obtained written informed consent form the infant's parents or legally authorized representatives (LAR).
4. Infant aged between 1 and 8 months.
5. Exclusively formula-fed at time of enrolment; or CMPA infant receiving partial breastfeeding and infant's mother having independently elected before enrolment to exclusively formula feed.
6. Infants with physician-diagnosed CMPA as per standard clinical practice:

Exclusion Criteria:

1. Previous treatment with AAF > 72 hours
2. Known underlying medical condition that would impair growth (as per physician's assessment, e.g. unstable congenital heart disease, cystic fibrosis, metabolic disorder, chronic liver disease etc.)
3. Demonstrated chronic malabsorption which is not due to CMPA.
4. Other significant pre-natal and/or serious post-natal disease other than CMPA before enrolment (per investigator's medical decision).
5. Infants whose parents or caregivers who cannot give informed consent or who cannot be expected to comply with study procedures.
6. Treatment with systemic corticosteroids (oral or intravenous) for >72 hours within 4 weeks before enrolment (topical corticosteroids allowed)
7. Infants taking probiotic preparations for > 72 hour within 4 weeks before enrolment
8. Currently participating or having participated in another clinical trial since birth.

Ages: 1 Month to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Full-term infants 1-8 months of age with symptoms suggestive of moderate-to-severe CMPA who have failed a trial of extensively hydrolyzed formula (EHF) of at least 2 weeks or who require amino acid formula as first line of treatment
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The weight-for-age z-score (WAZ) compared with the WHO 2006 Child Growth Standard | Comparison of baseline WAZ vs WAZ at 4 months
  Weight gain will be measured in kg and converted to WAZ scores

SECONDARY OUTCOMES:
Length-for-age Z-scores (LAZ) compared with the WHO 2006 Child Growth Standard | 1, 2, 3, 4 months from baseline and at 12 months of age
  Body length will be measured in cm and converted to LAZ scores

OTHER OUTCOMES:
Head circumference (HCAZ) compared with the WHO 2006 Child Growth Standard | 1, 2, 3, 4 months from baseline and at 12 months of age
  Head circumference will be measured in cm converted to HCAZ scores
Monitoring of CMPA-related symptoms | 1, 2, 3 and 4 months from baseline and at 12 months of age
  CMPA-related symptoms will be documented by the study physician on data collection forms
Faecal microbial composition | Enrolment,1, 2, 3 and 4 months from treatment start and also at 12 months of age
  Faecal samples will be collected before and after the study formula ingestion
Product compliance | 1, 2, 3 and 4 months from baseline and at 12 months of age
  Daily quantity consumed (mL) will be recorded for the 3 days preceding each visit in a diary given to the parent or caregiver

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital at Westmead, Sydney, Westmead, Australia